CLINICAL TRIAL: NCT05375045
Title: Real-life Evaluation of the Safety and Performance of EUROTEKNIKA Dental Implants
Status: Recruiting | Type: Observational
Sponsor: Euroteknika (Industry)
Collaborators: EVAMED (Other)
Responsible Party: Sponsor
Other Study IDs: SUIVI IMPLANTS
Record Dates: First submitted 2022-03-03; First posted 2022-05-16 (Actual); Last update posted 2022-05-16 (Actual); Status verified 2022-05

CONDITIONS: Edentulous Mouth
MeSH Terms: conditions — Mouth, Edentulous | interventions — Dental Implantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- prospective: A prospective cohort will be recruited into the study to meet the secondary objective of improving quality of life. In fact, to measure the improvement in quality of life, a questionnaire must be completed by the patient before the implant is placed. Answers to this questionnaire preoperatively cannot be collected for patients recruited retrospectively.
  Interventions: Device: dental implantation
- retrospective: Patients who received one or more EUROTEKNIKA implants before 2017 may be included in the study for the retrospective cohort

INTERVENTIONS:
Device: dental implantation — an implant is surgically inserted into the maxilla or mandible, and then an abutment is connected to this implant to support the dental prosthesis.
  Groups: prospective

SUMMARY:
Real-life evaluation of the safety and performance of EUROTEKNIKA dental implants

DETAILED DESCRIPTION:
Many adults have one or more missing teeth. The negative consequences of partial or total edentulousness are numerous at the level of the orofacial sphere :

* Edentulism generates a strong aesthetic deficit due to the lack of support of the tissues and the facial musculature;
* Edentulism causes a functional deficit that can have significant repercussions on the nutritional status of the affected subject;
* Edentulism is accompanied by bone resorption of the jaws which is unavoidable in the absence of implant treatment;
* In addition, the resulting feelings of discomfort and fragility are experienced as a real psychological handicap by the patient, partially or totally edentulous, which can then have significant repercussions on his social life.

EUROTEKNIKA dental implants are intended to be used for the replacement of a dental root in order to support a fixed or mobile prosthesis and thus restore masticatory function. EUROTEKNIKA dental implants are made of titanium or titanium alloy for surgical implants in accordance with ISO5832-2 and -3 standards.

EUROTEKNIKA dental implants are intended for use in cases of single, partial or complete edentulism on the maxillary and/or mandibular arch:

* Single tooth loss,
* Intercalary toothlessness,
* Terminal toothlessness,
* Total edentulism.

Dental implantology is based on the following principle: an implant is surgically inserted into the maxilla or mandible, and then a pillar is connected to this implant to support the dental prosthesis.

The use of dental implants is based on a biological process called osseointegration. Osseointegration corresponding to the fact that certain materials such as titanium are able to form direct contact with the surrounding bone. Osseointegration is therefore the direct structural and functional connection between living bone and the surface of an artificial implant. In order to allow the osseointegration process, and depending on the clinical case, a more or less long healing period must be observed before connecting the prosthetic elements to the implant. In cases of immediate loading, there is no healing period.

The expected benefits of this surgery are to improve the quality of life of patients and to recover masticatory function.

The claimed clinical performances are:

* High primary stability,
* High long-term implant stability,
* Limitation of bone resorption and risks of mucositis and peri-implantitis
* Maintenance of soft tissues.

The objectives of this study are therefore to assess the safety and performance of EUROTEKNIKA dental implants.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 or over
* Patient who has completed bone growth
* Patient informed and agreeing to participate in the study
* Partially or totally edentulous patient who will be implanted with the EUROTEKNIKA dental implant (for the prospective cohort)
* Patient to benefit from the placement of an implant for the creation of a single crown (for the prospective cohort)
* Patient implanted with the EUROTEKNIKA dental implant before 2017 (for the retrospective cohort)
* Patient having benefited from the placement of an implant for the creation of a single crown (for the retrospective cohort)

Exclusion Criteria:

* Pregnant or breastfeeding women (for the prospective cohort)
* Patient with bone disease in the cervico-facial region
* Patient refusing to participate in the study
* Patient with at least one contraindication to implantation (for the prospective cohort)
* Patient to benefit from the placement of an implant with immediate or early loading (for the prospective cohort)
* Patient to benefit from the placement of an implant for the support of the bridge, piles, attachment (for the prospective cohort)
* Patient having benefited from the placement of an implant with immediate or early loading (for the retrospective cohort)
* Patient having benefited from the placement of an implant for the support of the bridge, piles, attachment (for the retrospective cohort)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who received one or more EUROTEKNIKA implants before 2017 may be included in the study for the retrospective cohort for Naturactis, Naturall+, Aesthetica+2, ORIGIN, iBone E, iBone S and iBone G implants. These patients will be included consecutively in chronological order to avoid selection bias.
  A prospective cohort will also be recruited in the study, in order to meet the secondary objective concerning the improvement of the quality of life. In fact, to measure the improvement in quality of life, a questionnaire must be completed by the patient before the implant is placed. Answers to this questionnaire preoperatively cannot be collected for patients recruited retrospectively.
Sampling Method: Non-Probability Sample
Enrollment: 868 (Estimated)
Dates: Start 2022-03-25 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2028-02-01 (Estimated)

PRIMARY OUTCOMES:
The success rate of tissue integration of the implant | 5 years after implantation
  Integration of the implant 5 years after implantation

SECONDARY OUTCOMES:
assessment of the quality of life of patients following the recovery of full dentition with the GOHAI score (General Oral Health Assessment Index) | 5 years after implantation
  the quality of life of patients will be evaluated with the GOHAI score before implantation and 5 years after implantation
Complication rate taking into account pain, local tenderness, infection, mobility of the implant, fracture | 5 years after implantation
  pain, local tenderness, infection, mobility of the implant, fracture will be collected during the 5 years follow-up
measuring chewing function after prosthesis placement | 5 years after implantation
  Occlusal assessment will be performed after implantation and at 5 years follow-up
Rate of inflammation (visual) | 5 years after implantation
  Assessment of inflammation with visual examination 5 years after implantation
Assessment of the evolution of the péri-implant tissues | 5 years after implantation
  assessment of the evolution of the péri-implant tissues with the Pink esthetic score
assessment of the osseointegration of the implant | 5 years after implantation
  assessment of the osseointegration of the implant with the ISQ score
Rate of infection (x-ray) | 5 years after implantation
  Assessment of infection with radiographic examination 5 years after implantation

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Clermont Ferrand, Clermont-Ferrand, France

IPD SHARING:
Plan to Share IPD: No